CLINICAL TRIAL: NCT06520436
Title: Arthroscopic-Assisted Reduction for Developmental Dislocation of The Hip Through the Sub-Adductor and Anterolateral Portals
Brief Title: Arthroscopic-Assisted Reduction of Hip Dislocation Via Sub-Adductor and Anterolateral Portals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed El-Desouky, Associate Professor of Orthopedic surgery, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD-411-2018
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arthroscopic-Assisted Reduction (Experimental)
  Interventions: Procedure: Arthroscopic-Assisted Reduction

INTERVENTIONS:
Procedure: Arthroscopic-Assisted Reduction — The arthroscopic-assisted reduction was used as a one-stage operative treatment for all hips. In addition to that, Dega pelvic osteotomy and/or femoral shortening and varus derotation osteotomies were performed when necessary.

SUMMARY:
This study aims to present our arthroscopic-assisted surgical technique's reliability as a successful treatment for DDH, achieving reduction without the potential sequelae associated with open reduction techniques.

DETAILED DESCRIPTION:
Developmental dysplasia of the hip (DDH) encompasses a spectrum of pathological conditions including dislocation, subluxation, and deformities of the femoral head and acetabulum. The optimal surgical approach for DDH remains a subject of debate. The goal of successful treatment is achieving a stable concentric reduction and preventing future subluxation or dislocation.The aim of this study is to introduce the reliability of our arthroscopic-assisted surgical technique as a successful treatment for DDH that can achieve reduction with avoidance of sequelae which may be experienced following open reduction techniques.

ELIGIBILITY:
Inclusion Criteria:

- Patients with DDH in this study

Exclusion Criteria:

- Previous surgical treatment and those with teratologic or neuromuscular dislocations

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Acetabular index | 1 year
Severin radiographic grading | 1 year
Modified Severin clinical grading | 1 year
Postoperative complications | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rashwan AS, El-Desouky M, Elbarbary H, Madbouly MAE, Khedr A. Arthroscopic-assisted reduction for Developmental Hip Dysplasia (DDH) through the sub-adductor and anterolateral portals; A 24-month follow-up prospective descriptive study. BMC Musculoskelet Disord. 2025 Jan 8;26(1):27. doi: 10.1186/s12891-024-08234-y. PMID 39773255